CLINICAL TRIAL: NCT06861309
Title: Evaluation of Innovative Placental Imaging Techniques in Fetal Growth Restriction
Brief Title: Placental Imaging Techniques
Status: Recruiting | Type: Observational
Sponsor: Carilion Clinic (Other)
Collaborators: Virginia Polytechnic Institute and State University (Other)
Responsible Party: Sponsor
Other Study IDs: IRB-24-2156
Record Dates: First submitted 2025-02-18; First posted 2025-03-06 (Actual); Last update posted 2025-03-06 (Actual); Status verified 2025-03

CONDITIONS: Fetal Growth Restriction (FGR); Placental Insufficiency; Preeclampsia; Still Births; Pregnancy; Pregnancy Complications; Pregnancy Outcomes; Ultrasound
Keywords: Fetal Growth Restriction; FGR; Placental Imaging; Utero-Placental Insufficiency; Growth Restriction; Ultrasound; Pregnancy; Pregnancy Complications; Maternal Fetal Medicine; Ultrafast Power Doppler Imaging; Quantitative Ultrasound; uPDI; QUS; MFM; Stillbirth; Preeclampsia; Verasonics; Verasonics Vantage 256; Carilion Clinic; Virginia Tech
MeSH Terms: conditions — Fetal Growth Retardation; Placental Insufficiency; Pre-Eclampsia; Pregnancy Complications; Stillbirth

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: Yes

GROUPS / COHORTS (2):
- Fetal-Growth-Restricted (FGR) Pregnancies: Eligible subjects diagnosed by standard-of-care, growth ultrasound with a fetal-growth-restricted (FGR) pregnancy will be assigned to this arm. All study participants, regardless of arm, will receive a combine ultrafast power Doppler imaging (uPDI) / quantitative ultrasound (QUS) research exam with the Verasonics Vantage 256 (Verasonics, Inc, Kirkland, WA) every three weeks from their growth ultrasound until delivery.
  Interventions: Device: ultrafast power Doppler imaging (uPDI) / quantitative ultrasound (QUS)
- Normal-Fetal-Weight Pregnancies: Eligible subjects diagnosed by standard-of-care, growth ultrasound with a normal-fetal-weight/healthy pregnancy will be assigned to this arm. All study participants, regardless of arm, will receive a combine ultrafast power Doppler imaging (uPDI) / quantitative ultrasound (QUS) research exam with the Verasonics Vantage 256 (Verasonics, Inc, Kirkland, WA) every three weeks from their growth ultrasound until delivery.
  Interventions: Device: ultrafast power Doppler imaging (uPDI) / quantitative ultrasound (QUS)

INTERVENTIONS:
Device: ultrafast power Doppler imaging (uPDI) / quantitative ultrasound (QUS) — All study participants, regardless of arm, will receive a combine ultrafast power Doppler imaging (uPDI) / quantitative ultrasound (QUS) research exam with the Verasonics Vantage 256 (Verasonics, Inc, Kirkland, WA) every three weeks from their routine growth ultrasound until delivery.

SUMMARY:
The goal of this proof-of-concept, case-control, clinical trial is to evaluate the efficacy of using two newer ultrasound technologies, quantitative ultrasound (QUS) and ultrafast power Doppler imaging (uPDI), to evaluate the health of the placenta, visualize blood flow through the placental vasculature by color Doppler imaging in singleton pregnancies with and without fetal growth restriction (FGR).

* Our primary objective is to investigate the ability of using these ultrasound technologies to distinguish healthy pregnancies from those affected by FGR, a condition characterized by a fetal weight below the 10th percentile for the gestational age or abdominal circumference of the pregnancy.
* Secondary aims include longitudinal evaluation of differences in QUS and uPDI imaging over gestation and changes in these measures with evolution of utero-placental insufficiency including with the development of abnormal umbilical-artery Doppler testing, diagnosis of severe FGR, identification of stillbirth, and detection of preeclampsia or preterm birth.

Investigators will compare QUS/uPDI imaging and values in pregnancies determined to be healthy by approved, standard-of-care growth ultrasounds to those diagnosed with FGR.

Participants will receive research ultrasounds with the experimental Verasonics Vantage 256 system (Verasonics, Inc, Kirkland, WA) utilizing uPDI/QUS every three weeks following their routine growth ultrasound evaluation until delivery. Demographic, obstetric, and delivery-related information, as well as portions of subjects' past medical history will be utilized by researchers to further contextualize imaging and variables gathered during the research ultrasounds.

DETAILED DESCRIPTION:
Background: This study is a proof-of-concept, case-control exploration of quantitative ultrasound (QUS) and ultrafast power Doppler imaging (uPDI) imaging techniques, applied to the placenta to evaluate health of the placenta, blood flow visualized by colored doppler imaging in patients with and without FGR. Investigators will utilize the Verasonics Vantage 256 research ultrasound machine (Verasonics, Inc, Kirkland, WA) for this study, which is not FDA approved/experimental, along with a standard-of-care Phillips ultrasound machine which is FDA approved.

Use of QUS gained interest within the 1980s to evaluate the health of a range of tissues, from myocardial [heart muscle], to artery plaques, to breast masses, to bone density. More recently, there has been great interest in QUS for evaluation of fetal tissue health, including fetal liver and lung tissue, as well as placental tissue to gauge both gestational age as well as placental health. QUS imaging creates a number of values including an attenuation coefficient estimate (ACE), specified in decibels (dB) which is a measurement of the ultrasound waves' absorption and scattering as they move through human tissue. QUS also generates other values including a frequency-dependent attenuation value. These numerical estimates of absorption and scattering along with others provided by QUS are believed to change within the placenta with increased gestational age due to increasing deposition of collagen and fibrin, two types of connective fibers. Measures of absorption, scattering, and related tissue properties may also be altered in unhealthy versus healthy placental tissue. Thus, QUS is believed to have the potential to inform the clinician about placental health which may be affected by uteroplacental insufficiency predisposing to fetal growth restriction. Researchers will also investigate power Doppler imaging (uPDI), a newer ultrasound modality that uses an ultra-high frame rate and clutter filtering to increase the Doppler imaging sensitivity. Traditional Doppler ultrasound displays color onto the normally greyscale ultrasound where blood flow is seen by the machine. However, traditional ultrasound with Doppler has difficulty in detecting blood flow within smaller vessels, such as the smallest spiral arteries of the placenta which provide nutrient and gas exchange to the fetus. It is believed uPDI may be able to better visualize these small vessels and other small areas of slow blood flow or pooled blood within the placenta, providing more direct evaluation of placental tissue perfusion and health.

Procedure: Ultrasounds will be performed every 3 weeks until delivery for both cohorts following informed consent. The first ultrasound will take place within 1 week of enrollment to allow for the sonographer to be scheduled. Ultrasounds will be performed by trained MFM sonographers. Ultrasounds will take place within the Maternal Fetal Medicine suite of Carilion Clinic [102 Highland Ave, Roanoke, VA], in clinical exam rooms with dimmable lights and calming music to reduce patient stress. Upon entering the exam room, IRB-approved study team members and/or sonographers will introduce themselves by name and capacity, then ask the name and date of birth of the subject to verify subject identity against the research enrollment log and EMR. The purpose for the visit will be reiterated and the subject's wish to continue to participate in the research will be verified to ensure continued consent. Any questions the subject has will be answered to the subject's satisfaction. An agenda for the encounter will be set by the IRB-approved study team member or sonographer, so the patient knows what to generally expect and how long the visit will take. The subject will be seated in a reclined position and asked to raise the bottom portion of their shirt, while the sonographer drapes the patient according to standard clinical procedure. Ultrasound gel will be applied to the subject's abdomen and the sonographer will then begin the ultrasound using the machine's transducer [part held in sonographer's hand].

To begin, an ultrasound using a standard-of-care, Philips ultrasound machine will be used to first verify continued fetal viability and perform a basic anatomical survey to ensure continued eligibility for the subject's given cohort [either Case [FGR-positive] or Control [FGR-negative]]. These Philips ultrasound machines are located in each of the standard MFM exam rooms. Following this, the sonographer will transition to the research ultrasound machine for the rest of the visit.

Participants will have research ultrasounds performed of their placentas using a Verasonics Vantage 256 system (a popular research ultrasound platform used for human imaging under IRB approval). The gestational age of the fetus, estimated fetal weight in grams, and growth/weight percentile measurements for that gestational age will be recorded during the research visits. The placenta will be scanned at a central, peripheral, and 'mid-disc' region to acquire QUS and uPDI images with the Verasonics research ultrasound as well. Three measurements will be acquired at these locations. The Verasonics machine will be programmed to project B-mode (brightness mode) images for the sonographer at the time of the research ultrasound for confirmation of correct placental location. These B- or brightness mode images will project a 2-dimensional, greyscale image of the placenta (or fetus) to the sonographer to orient him/her to the location they are scanning and find the placenta. The machine will be programmed to display thermal index (TI) and mechanical index (MI) during all exams, which are derived estimates of the heat and pressure created by ultrasound waves' energy. These are displayed for safety and kept within International Society of Ultrasound of Obstetrics and Gynecology (ISUOG) guidelines. The Verasonics machine will be programmed with a "hard stop" not to exceed these limits. The energy exposure from Ultrasound has no known cumulative effect. Following the ultrasound procedure, the subject will be cleaned of ultrasound gel with a cloth and drapes removed. The subjects will be told of any changes noticed since the last visit to the growth or health of their baby or placenta. Incidental findings obtained during the research ultrasound will be shared with the subject's routine clinical provider and the patient by IRB-approved and qualified physicians on the research team. The PI will advise the participant's routine clinical provider that all results obtained with the research ultrasound should be validated using an FDA Approved ultrasound and standard of care ultrasound techniques.

Following all research ultrasound procedures during the visit, subjects will be given an opportunity to ask any further questions they wish and receive answers to their satisfaction. Printouts of their baby from the standard-of-care ultrasound machine will be provided to subjects. Subjects will then be led back out of the MFM suite to the front desk where they will be scheduled for their next research visit.

Participants will not be under the primary care of the research physicians. The research physicians will not be involved in decisions regarding the timing, method, or procedures used to terminate a pregnancy or determining the viability of a neonate.

Analysis: Researchers will evaluate QUS and uPDI images of the placentas. Researchers will evaluate which QUS parameters are most strongly associated with FGR diagnosis by comparing them to numbers obtained by QUS in normal estimated fetal growth pregnancies. Researchers will examine uPDI images in FGR pregnancies versus those obtained from normal growth weight pregnancies.

Secondary analysis: Researchers will perform multimodal analysis to determine whether these ultrasound modalities can distinguish between pregnancies with: A.) confirmed diseases deriving from a placental origin; B.) abnormal umbilical artery assessments, severe FGR, preeclampsia and stillbirth; C.) no complications.

ELIGIBILITY:
Inclusion Criteria:

* Normal-Fetal-Weight Pregnancies Arm: Patient at least 18 to 45 years of age at screening
* Normal-Fetal-Weight Pregnancies Arm: Non-anomalous, singleton gestation without suspected genetic disorders or growth abnormalities
* Normal-Fetal-Weight Pregnancies Arm: Low-risk aneuploidy screening, if performed
* Normal-Fetal-Weight Pregnancies Arm: Intention to deliver at Carilion Roanoke Memorial Hospital (CRMH) or Carilion New River Valley Medical Center (CNRVMC)
* Normal-Fetal-Weight Pregnancies Arm: Anatomical survey has been performed
* Normal-Fetal-Weight Pregnancies Arm: 18 - 26 weeks gestational age without concern for fetal growth restriction (FGR) in the mid-trimester
* Normal-Fetal-Weight Pregnancies Arm: No substantial risk factors for FGR:

  1. Prior small-for-gestational age child
  2. Prior FGR pregnancy
  3. Prior preeclampsia
  4. Prior gestational hypertension (HTN)
  5. Current hypertension (HTN)
  6. Current smoking or nicotine use
  7. Current cocaine use
  8. Current In-vitro fertilization (IVF) pregnancy
  9. Current known vascular disease
  10. Pre-existing diagnosis of lupus
  11. Pre-existing diagnosis of diabetes mellitus [type I, II]
  12. Pre-existing diagnosis of severe anemia (Hb ≥ 7.9 g/dL)
* Normal-Fetal-Weight Pregnancies Arm: Pregnancy without current fetal growth restriction (FGR) diagnosis
* Normal-Fetal-Weight Pregnancies Arm: Subject willing and able to provide informed consent Note: Verify that the most recent version of the ICF was used to consent the subject
* Fetal-Growth-Restricted (FGR) Pregnancies Arm: Patient at least 18 to 45 years of age at screening
* Fetal-Growth-Restricted (FGR) Pregnancies Arm: Non-anomalous, singleton gestation without suspected genetic disorders
* Fetal-Growth-Restricted (FGR) Pregnancies Arm: Low-risk aneuploidy screening, if performed
* Fetal-Growth-Restricted (FGR) Pregnancies Arm: Intention to deliver at Carilion Roanoke Memorial Hospital (CRMH) or Carilion New River Valley Medical Center (CNRVMC)
* Fetal-Growth-Restricted (FGR) Pregnancies Arm: Anatomical survey has been performed
* Fetal-Growth-Restricted (FGR) Pregnancies Arm: Pregnancy diagnosed with fetal growth restriction (FGR) by estimated fetal weight <10th centile or abdominal circumference measurements <10th centile
* Fetal-Growth-Restricted (FGR) Pregnancies Arm: Subject willing and able to provide informed consent Note: Verify that the most recent version of the ICF was used to consent the subject

Exclusion Criteria:

* Normal-Fetal-Weight Pregnancies Arm: Multiple gestations
* Normal-Fetal-Weight Pregnancies Arm: Known fetal anomaly affecting biometric measurements
* Normal-Fetal-Weight Pregnancies Arm: Suspected fetal genetic disorder(s)
* Normal-Fetal-Weight Pregnancies Arm: Suspected fetal infection(s)
* Normal-Fetal-Weight Pregnancies Arm: Non-English or Spanish-speaking
* Normal-Fetal-Weight Pregnancies Arm: Unstable housing or transportation
* Normal-Fetal-Weight Pregnancies Arm: Any other criterion which, in the clinical judgement of the investigator, would make the subject unsuitable for study enrollment.
* Fetal-Growth-Restricted (FGR) Pregnancies Arm: Multiple gestations
* Fetal-Growth-Restricted (FGR) Pregnancies Arm: Known fetal anomaly affecting biometric measurements
* Fetal-Growth-Restricted (FGR) Pregnancies Arm: Suspected fetal genetic disorder(s)
* Fetal-Growth-Restricted (FGR) Pregnancies Arm: Suspected fetal infection(s)
* Fetal-Growth-Restricted (FGR) Pregnancies Arm: Non-English or Spanish-speaking
* Fetal-Growth-Restricted (FGR) Pregnancies Arm: Unstable housing or transportation
* Fetal-Growth-Restricted (FGR) Pregnancies Arm: Any other criterion which, in the clinical judgement of the investigator, would make the subject unsuitable for study enrollment.

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: Pregnancies affected by FGR and Healthy Pregnancies
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2025-03 (Estimated); Primary Completion 2026-02 (Estimated); Study Completion 2026-02 (Estimated)

PRIMARY OUTCOMES:
Number of spiral arteries detected by ultrasound | 40 weeks
Velocity of spiral artery jets detected by ultrasound | 40 weeks
Speed of sound detected by Quantitative Ultrasound | 40 weeks

SECONDARY OUTCOMES:
Number of Participants with Abnormal Umbilical Artery Doppler Measurement | 40 week
Rate of Preeclampsia in Participants | 40 week
Rate of Stillbirth in Participants | 40 week

CONTACTS AND LOCATIONS:
Overall Officials: Megan D Whitham, MD, Principal Investigator — Carilion Clinic
Locations (1):
- Carilion Clinic Maternal Fetal Medicine, Roanoke, Virginia, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Slator P, Aughwane R, Cade G, Taylor D, David AL, Lewis R, Jauniaux E, Desjardins A, Salomon LJ, Millischer AE, Tsatsaris V, Rutherford M, Johnstone ED, Melbourne A; participants of the workshop. Placenta Imaging Workshop 2018 report: Multiscale and multimodal approaches. Placenta. 2019 Apr;79:78-82. doi: 10.1016/j.placenta.2018.10.010. Epub 2018 Oct 31. PMID 30396518
- [Background] Hernandez-Andrade E, Huntley ES, Bartal MF, Soto-Torres EE, Tirosh D, Jaiman S, Johnson A. Doppler evaluation of normal and abnormal placenta. Ultrasound Obstet Gynecol. 2022 Jul;60(1):28-41. doi: 10.1002/uog.24816. PMID 34806234
- [Background] Monier I, Ego A, Benachi A, Ancel PY, Goffinet F, Zeitlin J. Comparison of the Hadlock and INTERGROWTH formulas for calculating estimated fetal weight in a preterm population in France. Am J Obstet Gynecol. 2018 Nov;219(5):476.e1-476.e12. doi: 10.1016/j.ajog.2018.08.012. Epub 2018 Aug 14. PMID 30118693
- [Background] Blue NR, Beddow ME, Savabi M, Katukuri VR, Mozurkewich EL, Chao CR. A Comparison of Methods for the Diagnosis of Fetal Growth Restriction Between the Royal College of Obstetricians and Gynaecologists and the American College of Obstetricians and Gynecologists. Obstet Gynecol. 2018 May;131(5):835-841. doi: 10.1097/AOG.0000000000002564. PMID 29630011
- [Background] Huang L, Wang Y, Wang R, Wei X, He Q, Zheng C, Peng H, Luo J. High-Quality Ultrafast Power Doppler Imaging Based on Spatial Angular Coherence Factor. IEEE Trans Ultrason Ferroelectr Freq Control. 2023 May;70(5):378-392. doi: 10.1109/TUFFC.2023.3253257. Epub 2023 Apr 26. PMID 37028058
- [Background] Deeba F, Ma M, Pesteie M, Terry J, Pugash D, Hutcheon JA, Mayer C, Salcudean S, Rohling R. Attenuation Coefficient Estimation of Normal Placentas. Ultrasound Med Biol. 2019 May;45(5):1081-1093. doi: 10.1016/j.ultrasmedbio.2018.10.015. Epub 2019 Jan 23. PMID 30685076
- See also: Verasonics Vantage 256 System — https://verasonics.com/vantage-systems/
- See also: Carilion Clinic Maternal Fetal Medicine — https://www.carilionclinic.org/locations/carilion-clinic-maternal-fetal-medicine
- See also: The American College of Obstetrics and Gynecology - Ultrasound Exam FAQ for Patients — https://www.acog.org/womens-health/faqs/ultrasound-exams
- See also: ACOG Guidelines for Diagnostic Imaging During Pregnancy and Lactation — https://www.acog.org/clinical/clinical-guidance/committee-opinion/articles/2017/10/guidelines-for-diagnostic-imaging-during-pregnancy-and-lactation